CLINICAL TRIAL: NCT01824121
Title: Autologous Mesenchymal Stem Cell Therapy in Progressive Supranuclear Palsy: a Randomized, Double-blind, Controlled Clinical Trial
Brief Title: Clinical Trial to Evaluate Bone Marrow Stem Cell Therapy for PSP, a Rare Form of Parkinsonism
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 032011; 2011-004051-39 (EudraCT Number)
Record Dates: First submitted 2013-03-31; First posted 2013-04-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-03

CONDITIONS: Progressive Supranuclear Palsy
Keywords: Progressive Supranuclear palsy; stem cell therapy
MeSH Terms: conditions — Supranuclear Palsy, Progressive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- immediate stem cell therapy (Active Comparator): patients will undergo active intervention i.e. they will be given stem cell therapy immediately. After 6 months they will undergo a sham procedure.
  Interventions: Biological: stem cell therapy
- delayed stem cell therapy (Sham Comparator): patients allocated to delayed stem cell therapy will undergo a sham procedure (incannulation of the femoral vein and infusion of saline solution). They will receive stem cell therapy after 6 months
  Interventions: Biological: stem cell therapy

INTERVENTIONS:
Biological: stem cell therapy — Bone marrow will be collected from the iliac crest under local anesthesia. Mesenchymal Stem Cells (MSCs) will be isolated and cultivated in vitro. Patients will be catheterized and the MSCs will then be administered by intra-arterial route via the internal carotid artery and the vertebral artery that is largest in caliber, injecting small boluses manually through a microcatheter.

SUMMARY:
There is evidence suggesting that stem cells harvested from the bone marrow and transplanted into the brain may be effective in slowing down the progression of parkinsonism. Mesenchymal stem cells are able to produce growth factors that provide support to diseased nervous cells.

In this study mesenchymal stem cells will be harvested from the bone marrow, cultivated in a test tube so that they multiply and then infused into the arteries that supply blood to the brain in 20 patients suffering from a rare form of parkinsonism, Progressive Supranuclear Palsy. Each patient will undergo two infusions, one with the stem cells and one without, at an interval of 6 months. The sequence of the two infusions will be assigned randomly; patients and assessors will not know the sequence (double-blind). Patients will be followed-up for up to 1 year after the last infusion, with regular assessments to assess safety, efficacy on motor and cognitive functions, and effects on the brain by neuroimaging techniques.

The study has a preliminary phase with 5 patients all given stem cell therapy alone, designed to assess safety

ELIGIBILITY:
Inclusion Criteria:

diagnosis of 'probable Progressive Supranuclear Palsy - Richardson's disease subtype' according to current diagnostic criteria (Litvan et al. 1996 and 2003)

* age at onset at least 40 years;
* disease duration 12 months to 8 years;
* supranuclear ophthalmoplegia;
* postural instability or falls within 3 years from disease onset
* positive MRI for PSP criteria (Quattrone et al, 2008)
* Stable pharmacological treatment for at least 90 days
* Lack of response to chronic levodopa (at least 12-month treatment).
* Able to stand in upright posture without assistance for at least 30 seconds
* Written informed consent (including video taping)

Exclusion Criteria:

* Idiopathic Parkinson's disease;
* Cerebellar ataxia
* Symptomatic autonomic dysfunction
* Evidence of any other neurological disease that could explain signs;
* History of repeated strokes with stepwise progression of parkinsonian features;
* History of major stroke;
* Any history of severe or repeated head injury;
* A history of encephalitis;
* A history of neuroleptic use for a prolonged period of time or within the past 6 months;
* Street-drug related parkinsonism;
* Significant other neurological disease on CT-scan/MRI;
* Oculogyric crises;
* Major signs of corticobasal degeneration;
* Signs of Lewy body disease;
* Other life-threatening disease likely to interfere with the main outcome measure;
* Any clinically significant laboratory abnormality, with the exception of cholesterol, triglycerides and glucose;
* Renal failure (serum creatinine more than 300 mM/l);
* Transaminase elevation more than twice the upper limit of normal;
* Any concomitant disorder associated with bone marrow function impairment
* Any concomitant disorder that requires chronic treatment with immunosuppressors, anti-inflammatory agents, and/or growth factors
* dementia (MMSE < 24 according to Folstein 1975 or defined according to DSM-IV TR criteria)
* any other disorder that could interfere with the evaluation of treatment or that could make intra-arterial infusion inadvisable
* any other features that, according to the investigator, could reduce adherence to protocol procedures or prevent rapid access in case of emergency;
* women of child-bearing age
* participation in another clinical trial with experimental treatment in the last 30 days
* brain MRI evidence of severe vascular abnormalities, space-occupying lesions or normal pressure hydrocephalus

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
incidence of adverse events | one year
  incidence of adverse events collected by clinical monitoring and performing routine laboratory tests

SECONDARY OUTCOMES:
changes in brain images | one year
  change vs baseline in the striatal density of dopamine transporters in SPECT brain images and in the normalized regional cerebral flow / glucose metabolism in the gray matter in PET brain images after one year

OTHER OUTCOMES:
changes in motor function | one year
  changes vs baseline in total and motor UPDRS scores, Hoehn & Yahr staging, SEADL score, CGI and multifactorial movement analysis
changes in cognitive functions | one year
  changes vs baseline in MMSE score and in a series of neuropsychological measures (verbal comprehension, perceptual organization, immediate memory, delayed memory, word list recognition, language attention / concentration, visuospatial ability, processing speed, executive function)

CONTACTS AND LOCATIONS:
Overall Officials: Rosaria Giordano, MD, Principal Investigator — IRCCS Ca' Granda Ospedale Maggiore Policlinico
Locations (1):
- ICP Parkinson Institute, Milan, Italy

REFERENCES:
- [Derived] Giordano R, Canesi M, Isalberti M, Marfia G, Campanella R, Vincenti D, Cereda V, Ranghetti A, Palmisano C, Isaias IU, Benti R, Marotta G, Lazzari L, Montemurro T, Vigano M, Budelli S, Montelatici E, Lavazza C, Rivera-Ordaz A, Pezzoli G. Safety and Effectiveness of Cell Therapy in Neurodegenerative Diseases: Take-Home Messages From a Pilot Feasibility Phase I Study of Progressive Supranuclear Palsy. Front Neurosci. 2021 Oct 12;15:723227. doi: 10.3389/fnins.2021.723227. eCollection 2021. PMID 34712113
- [Derived] Canesi M, Giordano R, Lazzari L, Isalberti M, Isaias IU, Benti R, Rampini P, Marotta G, Colombo A, Cereda E, Dipaola M, Montemurro T, Vigano M, Budelli S, Montelatici E, Lavazza C, Cortelezzi A, Pezzoli G. Finding a new therapeutic approach for no-option Parkinsonisms: mesenchymal stromal cells for progressive supranuclear palsy. J Transl Med. 2016 May 10;14(1):127. doi: 10.1186/s12967-016-0880-2. PMID 27160012
- [Derived] Giordano R, Canesi M, Isalberti M, Isaias IU, Montemurro T, Vigano M, Montelatici E, Boldrin V, Benti R, Cortelezzi A, Fracchiolla N, Lazzari L, Pezzoli G. Autologous mesenchymal stem cell therapy for progressive supranuclear palsy: translation into a phase I controlled, randomized clinical study. J Transl Med. 2014 Jan 17;12:14. doi: 10.1186/1479-5876-12-14. PMID 24438512